CLINICAL TRIAL: NCT04014439
Title: Relationship Between Neutrophil to Lymphocyte Ratio and Prealbumin Serum Levels With Diaphragm Thickness in Critical Patients
Brief Title: Relationship Between NLR and Prealbumin Levels With Diaphragm Thickness
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rudyanto Sedono, Medical Staff, Indonesia University
Other Study IDs: IndonesiaUAnes037
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Inflammatory Response
Keywords: diaphragm thickness; neutrophil to lymphocyte ratio; mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Diaphragm: Diaphragm thickness is 2 mm or more
  Interventions: Diagnostic Test: Ratio of Neutrophil to Lymphocyte; Diagnostic Test: Level of Prealbumin Serum
- Thinning Diaphragm: Diaphragm thickness is less than 2 mm
  Interventions: Diagnostic Test: Ratio of Neutrophil to Lymphocyte; Diagnostic Test: Level of Prealbumin Serum

INTERVENTIONS:
Diagnostic Test: Ratio of Neutrophil to Lymphocyte — Each patient was examined for a blood sample of 6 ml of venous blood taken from the cubital vein using a vacuum tube without anticoagulants. Blood samples were centrifuged at a speed of 3500 rpm for 20 minutes. Samples are processed with abbott® devices, to obtain neutrophil and serum lymphocyte levels. Plasma samples are stored in the refrigerator -20 C. The patient's diaphragm thickness was measured on days 0, 3, 5 and then the measurement was compared. Diaphragm thickness was measured in patients using mechanical ventilation in intensive care rooms.
Diagnostic Test: Level of Prealbumin Serum — Each patient was examined for a blood sample of 6 ml of venous blood taken from the cubital vein using a vacuum tube without anticoagulants. Blood samples were centrifuged at a speed of 3500 rpm for 20 minutes. Samples are processed with abbott® devices, to obtain neutrophil and serum lymphocyte levels. Plasma samples are stored in the refrigerator -20 C. The patient's diaphragm thickness was measured on days 0, 3, 5 and then the measurement was compared. Diaphragm thickness was measured in patients using mechanical ventilation in intensive care rooms.

SUMMARY:
A study to find the relationship between neutrophil to lymphocyte ratio (NLR) with diaphragm thickness of critical patients in ICU.

DETAILED DESCRIPTION:
Weaning from ventilator sometimes can be failed and it happened due to several factors. One of the causes was Ventilator Induced Diaphragm Dysfunction (VIDD). This VIDD process occurred due to thinning process of the diaphragm thickness or decreased diaphragm muscle mass. The whole process happened due to inflammatory reaction that usually appeared on patients in Intensive Care Unit (ICU). Thus, this study was aimed to find the relationship between neutrophil to lymphocyte ratio (NLR) with diaphragm thickness of critical patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Critical patients treated in intensive care unit using mechanical ventilation from day 0.
* Patients are clinically predicted to be treated for more than 5 days (qSOFA and clinical assessment)

Exclusion Criteria:

* History of suffering from neuromuscular disease and or diaphragmatic malformations
* Used non-invasive ventilation before starting to use mechanical ventilation
* History of tracheostomy
* Patients admitted to ICU within 12 months before this study

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are treated in intensive care unit and using mechanical ventilation from Day 0 till Day 5. These patients will be checked for their diaphragm thickness, level of prealbumin serums, and ratio of neutrophil to lymphocyte.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Level of Prealbumin Serum | 5 days
Ratio of Neutrophil to Lymphocyte | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Rudyanto Sedono, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li C, Li X, Han H, Cui H, Wang G, Wang Z. Diaphragmatic ultrasonography for predicting ventilator weaning: A meta-analysis. Medicine (Baltimore). 2018 Jun;97(22):e10968. doi: 10.1097/MD.0000000000010968. PMID 29851847
- [Result] Flevari A, Lignos M, Konstantonis D, Armaganidis A. Diaphragmatic ultrasonography as an adjunct predictor tool of weaning success in patients with difficult and prolonged weaning. Minerva Anestesiol. 2016 Nov;82(11):1149-1157. Epub 2016 Jul 12. PMID 27407022
- [Result] Conti G, Montini L, Pennisi MA, Cavaliere F, Arcangeli A, Bocci MG, Proietti R, Antonelli M. A prospective, blinded evaluation of indexes proposed to predict weaning from mechanical ventilation. Intensive Care Med. 2004 May;30(5):830-6. doi: 10.1007/s00134-004-2230-8. Epub 2004 Mar 20. PMID 15127195
- [Result] Sellares J, Ferrer M, Cano E, Loureiro H, Valencia M, Torres A. Predictors of prolonged weaning and survival during ventilator weaning in a respiratory ICU. Intensive Care Med. 2011 May;37(5):775-84. doi: 10.1007/s00134-011-2179-3. Epub 2011 Mar 4. PMID 21373820
- [Result] Khan J, Harrison TB, Rich MM. Mechanisms of neuromuscular dysfunction in critical illness. Crit Care Clin. 2008 Jan;24(1):165-77, x. doi: 10.1016/j.ccc.2007.10.004. PMID 18241784